CLINICAL TRIAL: NCT03230409
Title: Impact of Nursing Interventions on Adherence to Treatment With Anti-tuberculosis Drugs in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sant Joan de Deu (Other)
Collaborators: Official Barcelona Nurses Association (COIB) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: PIC-68-13
Record Dates: First submitted 2017-07-21; First posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Tuberculosis
Keywords: Tuberculosis, Latent Tuberculosis Infection, Adherence, Nursing, Pediatrics, Public Health.
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1, Retrospective (No Intervention): Routine outpatient follow-up visits were scheduled as follows: (a) in patients receiving primary chemoprophylaxis or Latent Tuberculosis Infection (LTBI) treatment: baseline visit, and 2 weeks and 3 months later (end of treatment in most cases); (b) in patients treated for Tuberculosis disease: baseline visit, 2 weeks later and on a monthly basis thereafter.
- Phase 2, Prospective (Experimental): Four nurse-led interventions were implemented after Phase 1:
  * Intervention 1: at baseline visit, the parents or carers of the children, were given a leaflet in the mother tongue. This leaflet was available in 10 different languages: Spanish and Catalan (the two official languages of the country), English, French, German, Russian, Romanian, Chinese, Urdu and Arabic.
  * Intervention 2: a follow-up open telephone call was made 7-10 days after the baseline visit and whenever the patient failed to attend the scheduled visits.
  * Intervention 3: the Eidus-Hamilton test was performed twice, 2 weeks after the baseline visit and at the end of treatment. To prevent patients from only taking their medication occasionally, directly before their visits, they were not informed of the purpose of the urine test.
  * Intervention 4: a written questionnaire about adherence to anti-TB treatment on all the follow-up visits.
  Interventions: Behavioral: Leaflet written in the patient's/family mother tongue; Behavioral: A follow-up telephone call; Biological: Eidus-Hamilton Test; Behavioral: A written questionnaire

INTERVENTIONS:
Behavioral: Leaflet written in the patient's/family mother tongue — At baseline visit, the parents or carers of the children and/or the young patients themselves (in the case of adolescents >12 years of age), were given a leaflet including questions and answers about the most common doubts that people have about anti-TB treatment (what to do if you forget a dose, if you vomit, if you have stomach ache, etc.). The study nurse read and reviewed the leaflet with the family. This leaflet was available in 10 different languages: Spanish and Catalan (the two official languages of the country), English, French, German, Russian, Romanian, Chinese, Urdu and Arabic.
  Arms: Phase 2, Prospective
Behavioral: A follow-up telephone call — A follow-up open telephone call was made 7-10 days after the baseline visit and whenever the patient failed to attend the scheduled visits. The parents and/or patient were informed about this. This call was made to reinforce the information, answer any questions that may have arisen and insist on the importance of proper follow-up.
  Arms: Phase 2, Prospective
Biological: Eidus-Hamilton Test — E-H test was performed twice, 2 weeks after the baseline visit and at the end of treatment. To prevent patients from only taking their medication occasionally, directly before their visits, they were not informed of the purpose of the urine test. This test is a rapid, simple point-of-care method to detect urinary acetyl-isoniazid, the main metabolite of isoniazid, up to 12-24 hours following isoniazid administration and is used as a surrogate marker of treatment adherence. The test consists of placing 4 drops of a 10%potassium cyanide solution and 9 drops of a 10%chloramine solution in a test tube containing 4 drops of patient urine. The result is considered positive if a deep red color develops after 1 minute. If a pink color slowly appears,this indicates that there are only traces of the metabolite. If there is no change in color, the result is considered negative and suggests no recent isoniazid intake. The sensitivity and specificity of this test have been reported to be over 99%
  Arms: Phase 2, Prospective
Behavioral: A written questionnaire — The parents or carers of the children and/or the young patients themselves were asked to complete a written questionnaire about adherence to anti-TB treatment on all the follow-up visits, which was partially adapted from two validated questionnaires on adherence to chronic therapies (SMAQ compliance test, Svarstad et al., 1999; and Hermes test, Rodríguez-Chamorro et al., 2008).
  Arms: Phase 2, Prospective

SUMMARY:
This study evaluates the efficacy of nursing interventions on adherence to antituberculosis medication in a paediatric cohort (aged 0-18 years) and identifies the risk factors for non-compliance.

There are two phases in the study; Phase 1: retrospective descriptive analysis in children and young people receiving antituberculosis treatment (non-intervention group); and Phase 2: quasi-experimental, longitudinal, prospective study (intervention group). The results of the two phases will be compared.

DETAILED DESCRIPTION:
The study was carried out in the outpatient tuberculosis (TB) Unit of a tertiary-care pediatric center in Catalonia (Northeast Spain), which is a referral center for pediatric TB (Hospital Sant Joan de Déu) in the Southern Barcelona Health Care Region (Regió Sanitària Barcelona Sud) (1,346,000 inhabitants, 16.5% of whom are under 18 years of age).The TB incidence rate in Catalonia has decreased from 21.6 per 100,000 population in 2004 to 14.4 in 2015 (7.3 cases per 100,000 population of pediatric age)(Rodés, Espinilla, & García, 2016).

In both phases, all children and adolescents (aged <18 years) starting anti-tuberculosis (anti-TB) treatment due to close contact with a TB patient (primary chemoprophylaxis), Latent Tuberculosis Infection (LTBI) or TB disease were eligible to participate in the study. Directly Observed Treatment (DOT) is not routinely available in Spain, and its use is restricted to individual cases, as per physician decision.

The number of children and adolescents required to participate in the study was calculated using a unilateral chi-square proportion comparison test for independent samples, with a level of significance of 5% and a power of 80%, a 2/1 ratio in Phase 1/Phase 2 group sizes and assuming a significant increase of 15% in the adherence rate after the nurse-led interventions (60% in Phase 1 and 75% in Phase 2). Thus, it was calculated that 182 and 91 children and adolescents would be needed in the Phase 1 and Phase 2 groups, respectively.

Procedure and interventions:

As per national guidelines, primary chemoprophylaxis after TB contact consists of isoniazid in monotherapy until TB infection screening is repeated 10-12 weeks later. Treatment of LTBI includes either 3 months of isoniazid and rifampicin or 6-9 months of isoniazid in monotherapy, and treatment of TB disease consists of a 2-month induction phase with 4 drugs (isoniazid, rifampicin, pyrazinamide and ethambutol), followed by isoniazid and rifampicin for a minimum of 4 months.

Routine outpatient follow-up visits were scheduled as follows: (a) in patients receiving primary chemoprophylaxis or LTBI treatment: baseline visit, and 2 weeks and 3 months later (end of treatment in most cases); (b) in patients treated for TB disease: baseline visit, 2 weeks later and on a monthly basis thereafter.

Four nurse-led interventions were implemented after Phase 1: 2 educational interventions (leaflet in mother tongue and a follow-up open telephone call) and 2 monitoring interventions (the Eidus-Hamilton test and a written questionnaire about adherence to anti-TB treatment), which were exclusively carried out by 2 study nurses.

Whenever the Eidus-Hamilton test or the written questionnaire were consistent with sub-optimal adherence, immediate feedback was given to the parents and the patient the study nurse underlined the importance of adherence, assessed any potential hindrances and answered any questions. A follow-up visit or telephone call was scheduled 7-10 days later.

The level of adherence to anti-TB treatment was be identified retrospectively in Phase 1 of the study, as the risk factors associated with adherence in our cohort. Once Phase 2 was completed, the results were be compared with those of Phase 1 and the success of the new nurse-led interventions assessed.

Final results will be used to design the definitive Nurse-led Follow-up Programme that will be implemented in the TB Unit.

ELIGIBILITY:
Inclusion Criteria:

* In both phases, all children and adolescents (aged <18 years) starting anti-TB treatment due to close contact with a TB patient (primary chemoprophylaxis), Latent Tuberculosis Infectious (LTBI) or Tuberculosis (TB) disease were eligible to participate in the study.

Exclusion Criteria:

* Referral from another center after anti-TB treatment had already begun
* Patients with other chronic diseases requiring hospital follow-up and/or other chronic therapies
* Known poor previous adherence to anti-TB treatment (if treatment was repeated or restarted)
* A significant language barrier that prevented the child or his/her relatives from properly understanding the nature of the study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 359 (Actual)
Dates: Start 2014-01-01; Primary Completion 2016-09-30 (Actual); Study Completion 2017-01-15 (Actual)

PRIMARY OUTCOMES:
Adherence to treatment | Through the study completion, an average of 3 months for those patients starting anti-TB treatment due to close contact with a TB patient (primary chemoprophylaxis) or LTBI and 6-9 months for those with TB disease.
  Non-adherence was defined as the presence of any of the following situations:
  1. At the follow-up visits, it was calculated and/or the children or relatives stated that they had failed to take >20% of the previously prescribed anti-TB treatment.
  2. The child failed to attend two or more of the scheduled visits without justification.
  3. DOT was indicated for any reason.
  4. The child or relatives intentionally stopped the previously prescribed anti-TB treatment.
  5. The Eidus-Hamilton urine test was negative on one or more follow-up visits.
  6. The written questionnaire showed that compliance was below 80% of the prescribed anti-TB treatment.

SECONDARY OUTCOMES:
Risk Factors | Through the study completion, an average of 3 months for those patients starting anti-TB treatment due to close contact with a TB patient (primary chemoprophylaxis) or LTBI and 6-9 months for those with TB disease.
  To identify epidemiological, clinical or social markers that make it possible to predict good or poor adherence to anti-TB treatment in children and young people.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Maria Guix-Comellas, Professor, Principal Investigator — Univeristat de Barcelona

IPD SHARING:
Plan to Share IPD: Yes
The Study Protocol has been published in Journal of Advanced Nursing
Supporting Information: Study Protocol, ICF
Time Frame: It is always available.
Access Criteria: Guix-Comellas, E. M., Rozas-Quesada, L., Force-Sanmartín, E., Estrada-Masllorens, J. M., Galimany-Masclans, J., & Noguera-Julian, A. (2015). Influence of nursing interventions on adherence to treatment with antituberculosis drugs in children and young people: research protocol. Journal of Advanced Nursing, 71(9), 2189-99. http://doi.org/10.1111/jan.12656
URL: http://doi.org/10.1111/jan.12656

REFERENCES:
- [Background] Amlabu V, Mulligan C, Jele N, Evans A, Gray D, Zar HJ, McIlleron H, Smith P. Isoniazid/acetylisoniazid urine concentrations: markers of adherence to isoniazid preventive therapy in children. Int J Tuberc Lung Dis. 2014 May;18(5):528-30. doi: 10.5588/ijtld.13.0730. PMID 24903787
- [Background] Cass AD, Talavera GA, Gresham LS, Moser KS, Joy W. Structured behavioral intervention to increase children's adherence to treatment for latent tuberculosis infection. Int J Tuberc Lung Dis. 2005 Apr;9(4):415-20. PMID 15830747
- [Background] Chang SH, Eitzman SR, Nahid P, Finelli ML. Factors associated with failure to complete isoniazid therapy for latent tuberculosis infection in children and adolescents. J Infect Public Health. 2014 Mar-Apr;7(2):145-52. doi: 10.1016/j.jiph.2013.11.001. Epub 2013 Dec 19. PMID 24361084
- [Background] Cruz AT, Starke JR. Increasing adherence for latent tuberculosis infection therapy with health department-administered therapy. Pediatr Infect Dis J. 2012 Feb;31(2):193-5. doi: 10.1097/INF.0b013e318236984f. PMID 21979799
- [Background] Garfield S, Clifford S, Eliasson L, Barber N, Willson A. Suitability of measures of self-reported medication adherence for routine clinical use: a systematic review. BMC Med Res Methodol. 2011 Nov 3;11:149. doi: 10.1186/1471-2288-11-149. PMID 22050830
- [Background] Guix-Comellas EM, Rozas L, Velasco-Arnaiz E, Morin-Fraile V, Force-Sanmartin E, Noguera-Julian A. Adherence to Antituberculosis Drugs in Children and Adolescents in A Low-Endemic Setting: A Retrospective Series. Pediatr Infect Dis J. 2017 Jun;36(6):616-618. doi: 10.1097/INF.0000000000001508. PMID 28030525
- [Background] M'imunya JM, Kredo T, Volmink J. Patient education and counselling for promoting adherence to treatment for tuberculosis. Cochrane Database Syst Rev. 2012 May 16;2012(5):CD006591. doi: 10.1002/14651858.CD006591.pub2. PMID 22592714
- [Derived] Guix-Comellas EM, Rozas-Quesada L, Velasco-Arnaiz E, Ferres-Canals A, Estrada-Masllorens JM, Force-Sanmartin E, Noguera-Julian A. Impact of nursing interventions on adherence to treatment with antituberculosis drugs in children and young people: A nonrandomized controlled trial. J Adv Nurs. 2018 May 3. doi: 10.1111/jan.13692. Online ahead of print. PMID 29726024